CLINICAL TRIAL: NCT05512676
Title: Trabectedin (T) in Combination With Pegylated Liposomal Doxyrubicin (PLD) Compared to Cisplatin Hypersensitivity (CH) Treatment in Recurrent Ovarian Cancer Patients Allergic to Carboplatin
Brief Title: Trabectedin/Caelyx vs Cisplatin Hypersensitivity in Relapsed Ovarian Cancer Patients Allergic to Platinum
Acronym: TvsCH
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Principal Investigator, Torbjørn Paulsen, Senior Consultant, Oslo University Hospital
Other Study IDs: 2015/2167 REK sør-øst B
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Neoplasm; Chemotherapeutic Toxicity; Chemotherapy Effect; Chemotherapy-induced Neutropenia; Chemotherapy-induced Nausea and Vomiting
Keywords: Ovarian cancer; Pegylated Liposomal Doxorubicin; Trabectedin; Cisplatin hypersensitivity; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Vomiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, clinical study. Intention to include 40 patients (20 patients treated with trabectedin and 20 with cisplatin hypersensitivity) The investigators investigate the role of trabectedin in combination with PLD and cisplatin in treating platinum sensitive ROC being allergic to carboplatin. The investigators focus on adverse events and evaluate if these are tolerable for the patients and further evaluate the measurable treatment effect on the tumor burden.

DETAILED DESCRIPTION:
INTRODUCTION Trabectedin (Yondelis®) is a tetrahydroisoquinoline alkaloid that is produced synthetically. It acts by interfering with DNA transcription factors, DNA binding proteins, and DNA repair pathways. This results in cell cycle arrest and apoptosis. Trabectedin (T) probably causes DNA double-strand breaks. Trabectedin decreases the level of proangiogenic VEGF, CCL2, and interleucin-6 (IL-6) which indicate that trabectedin is cytotoxic with immune regulatory effects (1).

Since 2007 trabectedin mainly has been used in the treatment of soft tissue sarcomas (1). In meningioma trabectedin has been used in a murine model of ovarian cancer (2). A combined treatment of trabectedin and anti-PD1 antibody produces a synergic antitumor effect (3).

In a phase III international multicentre study the addition of trabectedin to pegylated liposomal doxyrubicin (PLD) (Caelyx) has shown to improve progression free survival and overall response rate compared to PLD alone in second-line treatment of recurrent ovarian cancer (ROC) (4). Trabectedin can replace platinum in clinical settings where there has been serious allergic reaction adverse effect from platinum (Carboplatin) (4). In many of these patients Carboplatin has been replaced by Cisplatin hypersensitivity regimen (CH). In patients with serious side effects to Cisplatin or other factors that impair the treatment of Cisplatin, trabectedin is a good alternative (4).

Trabectedin may also have a therapeutic role in patients with recurrent BRCA mutated ovarian cancer patients (5,6). When combined with PLD, trabectedin improves progression free survival (PFS) and objective response rate (ORR) in the second line-treatment of ROC. The combination led to manageable and non-cumulative overall toxicity with a fewer PLD-associated adverse events (7,8,9).

The majority of patients treated with trabectedin are given the combination with PDL and patients treated with cisplatin have the combination with paclitaxel.

In the present study the investigators will examine the role of trabectedin in combination with PLD and cisplatin in treating platinum sensitive ROC being allergic to carboplatin. The investigators will focus on adverse events and evaluate if these are tolerable for the patients and further evaluate the measurable treatment effect on the tumor burden.

Primary aims:

To investigate if trabectedin in combination with pegylated liposomal doxyrubicin (PLD) is applicable to replace desensitising cisplatin ROC treatment.

Secondary aims:

* Effect on tumor burden (CT by RISK criteria, vaginal ultrasound, CA125).
* Level of adverse effects.
* To calculate the PFS of the two cohorts (trabectedin and cisplatin).
* To calculate cancer specific survival (CSS) of the two cohorts (trabectedin and cisplatin) MATERIAL AND METHODS A description of the indication of treatment and follow-up after treatment with trabectedin in combination with PLD or cisplatin at the Oslo University Hospital (OUS), Department of gynecologic cancer. This study is retrospective and prospective in design. Totally 20 patients treated with trabectedin in combination with PLD and 20 patients with cisplatin will be included in the study.

Platinum sensitive tumors are defined as tumors recurring 6 months or more after previouis platinum treatment. In the study the investigators will mainly include patients having allergic reactions to carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Women with recurrent ovarian cancer and
* allergic reaction to carboplatin or
* other serious side effects to carboplatin

Exclusion Criteria:

- Patients not treated with carboplatin previously

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women included
Study Population: * Inclusion of 20 patients treated with trabectedin and pegylated liposomal doxorubicin after at least one line of previous chemotherapy.
  * Inclusion of 20 patients treated with cisplatin hypersensitivity and paclitaxel after at least one line of previous chemotherapy
  * All patients treated at Oslo University Hospital, Dept. Gyn. Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
PFS | From date of end of recurrent treatment (date of last cycle) with trabectedin/PLD or cisplatin hypersensitivity/paclitaxel until the date of first documented progression or date of death from any cause whichever came first, assessed up to 130 months.
  Progression Free Survival
Side effects | The side effects are assessed until 28 days after each cycle, up to 8 weeks after last cycle with trabectedin or cisplatin hypersensitivity. Each cycle is 28 days until 6 cycles..
  Side effects of recurrent treatment from trabectedin/PLD and cisplatin hypersensitivity/paclitaxel.

SECONDARY OUTCOMES:
Cancer Specific survival (CSS) | From date of primary diagnosis until date of last observation or death of ovarian cancer, whichever came first, assessed up to 36 years.
  Cancer Specific survival
Drug Interactions | From date of start recurrent treatment with trabectedin/PLD or cisplatin hypersensitivity/paclitaxel until date of last cycle with trabectedin/PLD or cisplatin hypersens/paclitaxel. The data are assessed at each cycle, 2 weeks after each cycle until 6.
  Interactions between trabectedin/PLD or cisplatin hypersensitivity/paclitaxel and other drugs the patients use during recurrent treatment (Examples: antihypertensive drugs, drugs inhibition of CYP450 2C8/3A4). The drugs are defined as mild increase-moderate increase -severe increase, mild decrease, modereate decrease, and severe decrease (6 categories) of trabectedin, PLD, cisplatin hypersensitivity or paclitaxel effect. The categories are obtained from the Drug Interactions Checker at www.drugs.com.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rokkones, PhD, Study Director — Head of Gyn. Onc. Department, Oslo University Hospital; Torbjørn Paulsen, PhD, Principal Investigator — Oslo University hospital, Dept. Gyn. Oncology, Norway

IPD SHARING:
Plan to Share IPD: Yes
The data are saved in individual Case Report Forms in pdf format. All data are encoded in SPSS. An anonymous SPSS File may be distributed on request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: End of 2023
Access Criteria: A description of the purpose of data sharing.